CLINICAL TRIAL: NCT04930380
Title: Description of Adherence to the Main Preventive Health Campaigns of Persons With Multiple Sclerosis
Acronym: preventionMS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Monica Ulivelli, principal investigator, University of Siena
Other Study IDs: 2021/Special-Multi/004
Record Dates: First submitted 2021-06-03; First posted 2021-06-18 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Multiple Sclerosis
Keywords: preventive medicine
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: * male and female aged 25 years or more
  * diagnosis of defined MS
  * written informed consent must be obtained before the enrolment.
  Interventions: Other: phone interview
- Controls: * male and female aged 25 years or more
  * written informed consent must be obtained before the enrolment no history of MS
  Interventions: Other: phone interview

INTERVENTIONS:
Other: phone interview — Cases and controls will receive a phone interview

SUMMARY:
Persons with multiple sclerosis (PwMS) might be more susceptible to infections and cancers and chronic diseases than general population, not because of the presence of the disease itself, but in relation to some specific therapies use or the degree of disability. Based on the currently available knowledge, the use of many disease-modifying drugs (DMDs) requires special attention to the possibility of infectious events or onset of cancer. In this perspective, a still unmet clinical need in PwMS is the acquisition of a complete picture of the immunization status against the main infectious diseases and the risk of cancer and other chronic diseases. Adherence to preventive pathways can reduce screening time for access to specific treatments, increase safety within complex therapies and reduce the risk of comorbidities.

Despite of the relevance of preventive medicine in clinical decision making, there are no studies in literature on the adherence of these patients to screening and vaccination campaigns in Italy.

The purpose of the study will be to describe the adherence to preventive medicine by PwMS, investigating possible differences between PwMS and people without MS (PwoMS) in the access to vaccinations and screenings. In addition, the investigators will try to identify, in both groups, the potential variables correlated to preventive medicine adherence, including the influence of the Covid(Coronavirus disease)-19 pandemic.

This 1-year project is conceived as a multicenter, observational and retrospective study, divided in two parts. The first one is conceived as a cross-sectional study that will enrol approximately 1250 patients from databases of Clinical Centers, Rehabilitation Units and local branches of the Italian MS Society in Northern, Central and Southern Italy. Patients over 25 years of age with a confirmed diagnosis of MS will be enrolled. Data will be collected through a questionnaire administered by telephone, upon written informed consent.

The second part is designed as a case-control study, that will enrol a subgroup of 300 PwMS (case group) and 300 PwoMS, matched by gender, age and residence area (control group) to analyse the impact of disease and/or disability to access/adherence to preventive medicine.

Knowledge of immunization status and chronic diseases risk is critical for clinical practice in the management of new DMDs but also for public health in determining the possible need for integrated care pathways targeted to PwMS.

DETAILED DESCRIPTION:
Disease prevention is a set of "specific, population-based and individual-based interventions for primary and secondary (early detection) prevention, aiming to minimize the burden of diseases and associated risk factors.". Depending on the objectives and the type of intervention, three levels of prevention are distinguished:

* "Primary prevention: intervening before health effects occur, through measures such as vaccinations, altering risky behaviours, and banning substances known to be associated with a disease or health condition"
* "Secondary prevention: screening to identify diseases in the earliest stages, before the onset of signs and symptoms"
* "Tertiary prevention: managing disease post diagnosis to slow or stop disease progression through measures" In this study the investigators will take in account primary prevention, including vaccine, tobacco smoke, alcohol consumption and body mass index, and secondary one, considering screening tests.

Primary prevention: Vaccine is a biological preparation that provides active acquired immunity to a particular pathogen and it represent "a simple, safe, and effective way of protecting people against harmful diseases, before they come into contact with them.". Vaccination "represent one of the most effective and cost-effective medical and public health achievements of all time" with the aim to protect not only the individuals but also the population. According to WHO (world health organization), "immunization is a key component of primary health care and an indisputable human right". In Italy there is a lifetime immunization schedule establishes the timing of mandatory and recommended vaccinations during all life.

Italian data on adult vaccination are available only for seasonal flu, reporting 15% of subjects vaccinated (53% >65, but only 9% in adults <64 even if with chronic diseases (22%)), and for rubella, showing that 39% of women of childbearing age are susceptible or unaware of their immune status.

Considering healthy lifestyle, most of Italian adults under 69 does not smoke (57%), but 18% is an ex-smoker and 25% smokes. Considering alcohol consumption, 44% of Italian adults does not consume alcohol, but 17% has a harmful use of it and 9% is a binge drinker. In addition, more than one-third of the Italian population aged 18 and over (35%) is in overweight, while just over one in ten is obese (11%).

Secondary prevention: Screening is defined as "the presumptive identification of unrecognized disease in an apparently healthy, asymptomatic population by means of tests, examinations or other procedures that can be applied rapidly and easily to the target population. A screening programme must include all the core components in the screening process from inviting the target population to accessing effective treatment for individuals diagnosed with disease". Mass screening involve the whole population, whereas the selective ones involve high-risk groups of population (but in certain cases they can be in large-scale, such as oncologic ones). Unlike diagnostic tests, used to make a diagnosis in symptomatic subjects, screening tests are aimed at asymptomatic but potentially at-risk people, indicating a suspicion of disease, and they can be repeated at regular interval.

Screening must be safe, simple and easy to administer, acceptable (with a minimal discomfort for subjects), inexpensive, reliable and valid, distinguishing diseased and non-diseased people. In Italy, organized screenings include tests for the detection of cervical, breast and colorectal cancer. In addition to these, family doctors (GPs) can control blood pressure and request diagnostic tests to control cholesterol, blood glucose, bone density and dermatological visits to check moles. The measurement of prostate antigen levels is another preventive investigation but is not currently considered a true screening because its usefulness is still a topic of discussion because PSA (prostatic specific antigen) screening could have more risks than benefits, especially. For this reason, the National centre for screening monitoring (ONS) does not recommend population PSA screening, and it recommends the test for diagnostic and non-preventive purposes only, especially for men>70.

In Italy, organized screening campaigns, the only ones monitored by the ONS and by Italian Behavioural Risk Factor Surveillance System (PASSI), have an adhesion rate varying according to geographical area. While coverage is almost complete in the Centre and the North, it remains insufficient in the South due to the smaller extension of organized programs and to the lower participation by citizens even with programs active. The coverage of mammography screening, recommended for women between 50 and 69 ys (in some Regions extended also to the age groups 45-49 and 70-74), reached 84% in the North, but only 62% in the South, although an increase was recorded also in this area. Cervical screening, recommended for women between 25 and 64 ys, reached 88% in the North, and 69% in the South. The coverage of colorectal screening, recommended for both sexes between 50 and 69 ys (in some Regions extended up to 74 ys), reached 69% in the North, while in the South still remained <28%.

In addition, other variables can also affect the adherence to screening campaigns, such as nationality, level of education and economic difficulties.

Moreover, the investigators have to consider that in the first 5 months of 2020, due to pandemic of Covid-19, ONS registered a decrease of more than one million of screening exams than the previous year.

Preventive medicine among people with multiple sclerosis/disabilities: Studies in the USA report a reduced access to preventive medicine for people with PwMS, especially for those with severe disabilities. Studies on unhealthy lifestyle in PwMS report a higher prevalence of smokers in PwMS than in general population, whereas for alcohol literature studies published discordant results. Regarding BMI, a recent American case control study report no difference on prevalence of overweight or obesity among PwMS and controls.

For Italy, however, there are no available study, and the American healthcare system differs greatly from the Italian one (mainly private vs public).

Regarding access to preventive medicine for subjects with various types of disabilities, the Italian Health Observation Report analysed adherence to mammography, pap-test, colorectal and flu vaccination campaigns (only for people over 65). The analysis showed that the number of women with functional limitations who perform mammography and pap tests is reduced by more than 15 percentage points than the general population. Regarding colorectal screening, men with disabilities show no difference compared to the general population, while disabled women adhere to the screening with a lower percentage.

Regarding the access to vaccinations, the one against influenza appears to be carried out by a higher percentage of men with disabilities than the Italian general population, but the study presents the bias of having a different demographic composition in the two considered cohorts since the one with functional limitation had more elders, for whom vaccination is more recommended. Also American studies report conflicting results: Diab et al. showed higher pneumococcal and seasonal flu vaccination rates in subjects with mild or medium disabilities compared to those without disabilities or with severe disabilities, while a previous study had found no difference between people with disabilities and the general population although both vaccinations are more recommended in people with disabilities or chronic diseases due to the greater risk of complications following infection.

Rationale and specific aims MS by itself do not increase the risk of other diseases, such as cancer, cardiovascular or infectious ones. Although the risk of infection associated with disability as well as the use of DMDs is well known, as well as their potential role in causing cancer disease as an adverse event.

This treatment scenario, with the increase in available DMDs in recent years, requires particular attention to tumour and infectious diseases both in the screening for therapy and follow-up. This could improve the adherence to screening campaigns due to a specific request of the neurologist.

Regarding the adherence to screening, it should be considered that PwMS with disabilities might have difficulties to access to preventive medicine due to functional limitations.

In Italy there are no specific studies on PwMS, although knowing the prevalence of patients who adhere to preventive medicine campaigns can be of great interest in public health decision-making, to launch eventual ad hoc preventive pathways for these subjects. In addition, having this information could help neurologists improving quality and timing in decision making for treatment selection. Adherence to preventive pathways can reduce screening time for access to specific treatments, increase safety within complex therapies and reduce the risk of comorbidities.

The Italian National Health Service guarantees integrated care pathways to people with complex needs, and Tuscany, have set up care pathways for people with a severe disability or special needs to promote fair access to health services, including prevention. This pathway could be set up, if necessary, specifically for PwMS, in synergy with the neurologists of the MS Centres and GPs who can play a strategic role in this area.

The purpose of the study will be to describe the adherence to preventive medicine by PwMS, investigating if there are differences between PwMS and people without MS (PwoMS) in the access to vaccinations and screenings. In addition, the investigators will try to identify, in both groups, the potential variables correlated to preventive medicine adherence, including the influence of the Covid-19 pandemic.

Considering that at 18 years of age the subjects have already received the mandatory and recommended vaccines provided by the vaccine calendar for childhood and adolescence, and that the first institutional screening campaign (pap-test) starts from 25 years of age, the latter was considered as the minimum age of enrolment in the study.

The enrolment of patients will be carried out on all macro-areas considered by the ONS in order to take into account the geographical differences present on the Italian Country. As previously mentioned, in fact, the coverage of screening campaigns and the adherence to them is lower in the South than in Central and Northern Italy.

The study will be carried out in two phases. A first phase consisting in a cross-sectional study to describe the adherence to medicine preventive of PwMS and a second phase, where a case-control study will be used to investigate differences in preventive medicine adherence between PwMS and PwoMS.

Phase 1 - Cross-sectional study Aim The specific aim will be to describe the adherence to medicine preventive of PwMS. Moreover, the investigators will evaluate variables which could affect the adherence to preventive medicine (screening and vaccines), such as sex, age, residence, nationality, education level, occupation, socio-economic status, quality of life, lifestyle (alcohol, smoke and BMI), MS forms, degree of MS-related disability and presence of chronic comorbidities. The possible impact of the ongoing Covid-19 pandemic will also be explored.

Phase 2 - Case-Control study Aim The specific aim will be to evaluate compliance rates for main screening tests and vaccines between PwMS and PwoMS and to investigate any differences in preventive medicine adherence between 2 groups. The investigators will use the same variables considered in the first phase of the study to evaluate the real impact of MS and disability level in the access/adherence of preventive measures, controlling for potentially confounding factors.

RESEARCH PLAN AND METHODS

Phase 1 - Cross-sectional study

Methods

Design and sample The study design will be a multicentric cross-sectional. Participants will be recruited in the study among PwMS attending the medium-large sized MS clinical centres, rehabilitation units or among PwMS in contact with the Italian Multiple Sclerosis Association (AISM). In the first two cases the subjects will be enrolled consecutively during ambulatory activities and in the third case the subjects will be randomly selected from the list of AISM's members. Healthcare workers/research assistants, trained for the purpose, will present the project to patients during enrolment. Subjects who give their consent to participate will be contacted by research assistants for a phone interview.

Data collection Subjects will complete an anonymous questionnaire combining socio-demographic, clinical and medicine preventive-related information and three scales validated in Italian, as described above. Two questionnaire form will be developed to take in account the sex difference (i.e. specific preventive screening such as mammography or prostate screening).

In particular, collected data will be:

* self-reported socio-demographic characteristics: age, sex, citizenship (if the interviewees are not Italian, the investigators will ask when they moved to Italy), province of birth, province of residence, level of education, marital status, employment status, income;
* self-reported clinical characteristics and lifestyle: year of onset and diagnosis of MS, type of course, presence of comorbidities, BMI, smoking and drinking use;
* self-reported preventive medicine-related information: main health screening (mammography and cervical screening -only for women-, colorectal screening, control of moles, blood pressure, cholesterol and blood sugar levels, bone density); main vaccines (dose booster of diphtheria/tetanus or diphtheria/tetanus/pertussis, the flu vaccine, the immunization status against rubella and chickenpox, the vaccine against HPV (Human papillomavirus, hepatitis B, meningococcus B, C and ACYW135, measles, pneumococcus and Herpes Zoster);
* level of disability: Self-Expanded Disability Status Scale (self-EDSS) will be used to measure subjects' level of disability. It is a descriptive scale derived from the original EDSS and also from the patient-assessed Patient Determined Disease Steps (PDDS). A recent evaluation of the feasibility and reliability of self-assessed EDSS has found it acceptable;
* level of independence in daily activities: Activities of Daily Living (ADL) Katz scale measures the ability of an individual to perform activities required in daily living. ADL scale consists of following six items: (1) bathing, (2) dressing, (3) transferring, (4) going to the toilet, (5) continence and (6) feeding. The total Katz ADL score indicates the degree of dependency. The range of the total score per item level is 1-4, with higher scores indicating a higher level of dependency: (1) independent, (2) requires some assistance, (3) requires full assistance and (4) completely dependent.
* quality of life: Eq-5D-3L will be used to measure the quality of life. The EQ(EuroQol)-5D-3L consists of two sections. In the first part, the descriptive system includes five single item dimensions of health (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). Each dimension is measured on a 3-point scale, and a single weighted score -the utility index- is obtained from these five questions. This score lies on a scale in which full health has a value of 1 and death has a value of 0, although negative values are allowed.

In addition, specific questions will ask if the MS disease or pandemic impact on access on preventive medicine.

Ethical considerations

Informed consent Eligible subjects will consent to participate after reading information about the study and what participation would entail and after providing written informed consent, by personally signing and dating the document. It will not be possible to proceed with the compilation of the questionnaire if consent is not provided.

Confidentiality The participation in the study is anonymous. The investigators must assure anonymity to enrolled subjects. For this reason, the documents sent to the coordinating Centre will be associated only with a number code identifying the patient and a letter code identifying the Center. However, the investigators of each Center must archive the listing of the identities of patients involved in the study.

Statistical methods Calculation of the sample size

The sample size calculation will be based on the prevalence of colorectal screening. A sample size will be estimated to ensure the recruitment of a sufficiently large number of participants stratified by geographical areas, to obtain statistically significant data. Assuming that the prevalence of colorectal screening in MS population is similar to that observed in a disable population given the chosen of margin error (5%), confidence interval (95%), assuming a 20% drop-out rate, it will be necessary an approximate population size of 1250 individuals. In particular sample size will consist of 460 persons resident in North, 460 in Centre and 330 in South Italy.

Analysis Descriptive statistics including means, frequencies and percentages will be used to analyze data. Frequencies will be used to describe screenings and/or vaccinations performed. To evaluate the variables correlated to probability to carry out preventive medicine, Chi-square and Fisher's exact tests will be used to assess for significance between categorical variables, whereas continuous ones will be analyzed using independent t-tests and ANOVA. Independent variables, resulting as significant (p <0.20) in the univariate analyses, will be included in multivariate models to determine the association between potential predictors and preventive medicine related outcomes (screening or vaccines). Preventive medicine related outcome will be dichotomized taking the value of 1 for receipt of the service and 0 for not having received the service. Separate multivariate logistic regression models will be built to generate odds ratios (ORs) and 95% confidence intervals (CIs) for each preventive health service.

. Phase 2 - Case-Control study (phase 1)

Methods

Design and sample The study design will be a multicentric matched case-control study (phase 1). The case and control subjects will be 1:1 matched to age, sex and residence area.

Case subjects will be PwMS enrolled consecutively among the subjects participating in phase 1 of the study.

Control subjects will be PwoMS volunteers. Control subjects will be enrolled among friends or neighbours of the cases. According to DL 15.07.1997, art 1.61, the enrolment of controls will not include vulnerable subjects, whose decision to volunteer in this project may be improperly influenced by the expectation, whether justified or not, of benefits associated with participation, or of possible retaliatory action by hierarchically superior individuals if they refuse to participate. Examples include members of hierarchically structured groups, such as medical, pharmacy, dental or nursing school students, subordinate hospital and laboratory staff, employees of a pharmaceutical industry, members of the armed forces, and prisoners. Other vulnerable individuals may include: patients with incurable diseases, persons housed in nursing homes, indigent persons, patients in emergency situations, ethnic minorities, homeless persons, nomads, refugees, minors, and persons incapable of giving consent. In addition, according to DL 24.0.2003 n 211, art 1, it is forbidden to offer, give or request financial incentives or benefits for the participation of the subjects in the study.

Data collection Control subjects will complete the same anonymous questionnaire combining socio-demographic, clinical (i.e. presence of comorbidity), lifestyle and medicine preventive-related information and some validated scales in Italian (see section Data collection in Phase 1 of the protocol).

In the same way as the cases, data regarding control subjects will be collected using a questionnaire that will completed during a telephone interview conducted by a research assistant trained ad hoc for the purpose.

Ethical considerations Informed consent Eligible case and control subjects may only be included in the study after providing written informed consent, by personally signing and dating the written informed consent document. Informed consent must be obtained before any data collection. In particular, case patient's willingness to participate upon informed consent will be subsequently followed by a request for names and contact information of two friends/neighbours. Control subjects have to be similar in age (within 5 years), sex and city of residence to the case patient. Case patients will be asked to contact their respective controls first and then to provide the potential controls' name and contact information once the potential control will have given their permission in study participation. The investigators will attempt to recruit and interview each friend/neighbour for whom the investigators will obtain contact information and written informed consent.

Confidentiality The participation in the study is anonymous. The investigators must assure anonymity to enrolled subjects. For this reason, the documents sent to the coordinating Centre will be associated only with a number code identifying the patient and a letter code identifying the Center. However, the investigators of each Center must archive the listing of the identities of patients involved in the study. Controls' questionnaire will have the same case code followed by the letter C.

Statistical methods Calculation of the sample size For the case-control study, the sample size will be calculated using the method described by Dupont. The sample size will be calculated with a power of 80% and two-sided confidence level of 95%. The expected compliance rates for screening of colorectal cancer will be considered as approximately 45% and 33% respectively in control and case group. The sample size was calculated to detect a minimum OR of 0.60. For a matched case-control study at a case to control ratio of 1:1, the required sample size will be 256 pairs of cases and controls. Assuming a 15% drop-out rate, 300 cases and 300 matched controls will be enrolled.

Analysis Descriptive statistics including means, frequencies and percentages will be used to analyze the data. Success of matching will be tested by comparing data between groups. For this purpose and to identify differences between groups in medicine preventive-related data, tests for matched pairs were used. Paired t- or Wilcoxon signed rank sum test (as appropriate) will be used for continuous data, while McNemar's or the Stuart-Maxwell test (as appropriate) for categorical data. Multivariable conditional logistic regression models, controlling for potentially confounding factors, will be used to compare preventive medicine adherence between the two groups.

All statistical tests will be 2-sided, and p<0.05 will be considered statistically significant. Analyses will be performed using Stata software, Version 15 (Stata Corp, College Station, Texas).

ELIGIBILITY:
Inclusion Criteria of cases:

* male and female aged 25 years or more
* written informed consent must be obtained before the enrolment
* diagnosis of defined MS

Exclusion Criteria of cases:

* under the age of 25
* unable to provide informed consent or to fill in the questionnaire

Inclusion Criteria of controls:

* male and female aged 25 years or more
* written informed consent must be obtained before the enrolment

Exclusion Criteria of controls:

* under the age of 25
* unable to provide informed consent or to fill in the questionnaire
* history of MS

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited in the study among PwMS attending the medium-large sized MS clinical centres, rehabilitation units or among PwMS in contact with the Italian Multiple Sclerosis Association (AISM). In the first two cases the subjects will be enrolled consecutively during ambulatory activities and in the third case the subjects will be randomly selected from the list of AISM's members. Healthcare workers/research assistants, trained for the purpose, will present the project to patients during enrolment. Subjects who give their consent to participate will be contacted by research assistants for a phone interview.
  Control subjects will be PwoMS volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 1250 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
questionnaire | 1 year
  adherence to preventive medicine

CONTACTS AND LOCATIONS:
Locations (12):
- Italy (12):
  - University of Ferrara, Ferrara, FE
  - University of Siena, Sena, SI
  - AOU San Luigi Gonzaga, Orbassano, TO
  - Aulss3- Ospedale dell'Angelo, Mestre, VE
  - Università di Cagliari, Cagliari
  - Università di Catania, Catania
  - Ospedale Murri, Fermo
  - Fondazione Italiana Sclerosi Multipla, Genova
  - Università degli Studi di Milano Statale, Milan
  - Università degli Studi di Palermo, Palermo
  - IRCCS Neuromed, Pozzilli
  - Università La Sapienza, Roma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shaw AR, Feinberg MB. Vaccines. Clinical Immunology. 2008;1353-1382. doi:10.1016/B978-0-323-04404-2.10092-2
- [Background] Hayes JH, Barry MJ. Screening for prostate cancer with the prostate-specific antigen test: a review of current evidence. JAMA. 2014 Mar 19;311(11):1143-9. doi: 10.1001/jama.2014.2085. PMID 24643604
- [Background] Barrett MW, Roberts B. Preventive Screening in People with Multiple Sclerosis. Int J MS Care. 2010;12:168-176.
- [Background] Dobos K, Healy B, Houtchens M. Access to Preventive Health Care in Severely Disabled Women with Multiple Sclerosis. Int J MS Care. 2015 Jul-Aug;17(4):200-5. doi: 10.7224/1537-2073.2013-046. PMID 26300706
- [Background] Bisson EJ, Ekuma O, Marrie RA, Leslie WD, Finlayson ML. Factors associated with receiving bone mineral density screening among people with multiple sclerosis. Mult Scler Relat Disord. 2019 Feb;28:305-308. doi: 10.1016/j.msard.2019.01.022. Epub 2019 Jan 8. PMID 30641355
- [Background] Shabas D, Weinreb H. Preventive healthcare in women with multiple sclerosis. J Womens Health Gend Based Med. 2000 May;9(4):389-95. doi: 10.1089/15246090050020709. PMID 10868611
- [Background] Beier M, D'Orio V, Spat J, Shuman M, Foley FW. Alcohol and substance use in multiple sclerosis. J Neurol Sci. 2014 Mar 15;338(1-2):122-7. doi: 10.1016/j.jns.2013.12.029. Epub 2013 Dec 27. PMID 24411661
- [Background] Russell RD, Langer-Gould A, Gonzales EG, Smith JB, Brennan V, Pereira G, Lucas RM, Begley A, Black LJ. Obesity, dieting, and multiple sclerosis. Mult Scler Relat Disord. 2020 Apr;39:101889. doi: 10.1016/j.msard.2019.101889. Epub 2019 Dec 9. PMID 31838309
- [Background] Diab ME, Johnston MV. Relationships between level of disability and receipt of preventive health services. Arch Phys Med Rehabil. 2004 May;85(5):749-57. doi: 10.1016/j.apmr.2003.06.028. PMID 15129399
- [Background] Iezzoni LI, McCarthy EP, Davis RB, Siebens H. Mobility impairments and use of screening and preventive services. Am J Public Health. 2000 Jun;90(6):955-61. doi: 10.2105/ajph.90.6.955. PMID 10846515
- [Background] Farez MF, Correale J, Armstrong MJ, Rae-Grant A, Gloss D, Donley D, Holler-Managan Y, Kachuck NJ, Jeffery D, Beilman M, Gronseth G, Michelson D, Lee E, Cox J, Getchius T, Sejvar J, Narayanaswami P. Practice guideline update summary: Vaccine-preventable infections and immunization in multiple sclerosis: Report of the Guideline Development, Dissemination, and Implementation Subcommittee of the American Academy of Neurology. Neurology. 2019 Sep 24;93(13):584-594. doi: 10.1212/WNL.0000000000008157. Epub 2019 Aug 28. PMID 31462584
- [Background] Riva A, Barcella V, Benatti SV, Capobianco M, Capra R, Cinque P, Comi G, Fasolo MM, Franzetti F, Galli M, Gerevini S, Meroni L, Origoni M, Prosperini L, Puoti M, Scarpazza C, Tortorella C, Zaffaroni M, Moiola L. Vaccinations in patients with multiple sclerosis: A Delphi consensus statement. Mult Scler. 2021 Mar;27(3):347-359. doi: 10.1177/1352458520952310. Epub 2020 Sep 17. PMID 32940128
- [Background] Lebrun C, Vukusic S; French Group for Recommendations in Multiple Sclerosis (France4MS) and the Societe Francophone de la Sclerose En Plaques (SFSEP). Immunization and multiple sclerosis: Recommendations from the French multiple sclerosis society. Mult Scler Relat Disord. 2019 Jun;31:173-188. doi: 10.1016/j.msard.2019.04.004. Epub 2019 Apr 10. PMID 31159998
- [Background] Melamed E, Lee MW. Multiple Sclerosis and Cancer: The Ying-Yang Effect of Disease Modifying Therapies. Front Immunol. 2020 Jan 10;10:2954. doi: 10.3389/fimmu.2019.02954. eCollection 2019. PMID 31998289
- [Background] Kurtzke JF. Rating neurologic impairment in multiple sclerosis: an expanded disability status scale (EDSS). Neurology. 1983 Nov;33(11):1444-52. doi: 10.1212/wnl.33.11.1444. PMID 6685237
- [Background] Hohol MJ, Orav EJ, Weiner HL. Disease steps in multiple sclerosis: a simple approach to evaluate disease progression. Neurology. 1995 Feb;45(2):251-5. doi: 10.1212/wnl.45.2.251. PMID 7854521
- [Background] Collins CD, Ivry B, Bowen JD, Cheng EM, Dobson R, Goodin DS, Lechner-Scott J, Kappos L, Galea I. A comparative analysis of Patient-Reported Expanded Disability Status Scale tools. Mult Scler. 2016 Sep;22(10):1349-58. doi: 10.1177/1352458515616205. Epub 2015 Nov 12. PMID 26564998
- [Background] Katz S, Akpom CA. A measure of primary sociobiological functions. Int J Health Serv. 1976;6(3):493-508. doi: 10.2190/UURL-2RYU-WRYD-EY3K. PMID 133997
- [Background] KATZ S, FORD AB, MOSKOWITZ RW, JACKSON BA, JAFFE MW. STUDIES OF ILLNESS IN THE AGED. THE INDEX OF ADL: A STANDARDIZED MEASURE OF BIOLOGICAL AND PSYCHOSOCIAL FUNCTION. JAMA. 1963 Sep 21;185:914-9. doi: 10.1001/jama.1963.03060120024016. No abstract available. PMID 14044222
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Naing L, Winn T, Rusli BN. Practical issues in calculating the sample size for prevalence studies. Arch Orofacial Sci 2006;1:9-14.
- [Background] Dupont WD. Power calculations for matched case-control studies. Biometrics. 1988 Dec;44(4):1157-68. PMID 3233252
- See also: Related Info — http://www.emro.who.int/about-who/public-health-functions/health-promotion-disease-prevention.html
- See also: Related Info — http://www.salute.gov.it/portale/influenza/dettaglioContenutiInfluenza.jsp?lingua=italiano&id=679&area=influenza&menu=vuoto
- See also: Related Info — https://www.epicentro.iss.it/passi/infoPassi/infoGen
- See also: Related Info — http://www.salute.gov.it/portale/documentazione/p6_2_2_1.jsp?lingua=italiano&id=1383
- See also: Related Info — https://www.osservatorionazionalescreening.it/sites/default/files/allegati/Rapporto_ripartenza-maggio_2020_def_0.pdf
- See also: Related Info — https://www.gov.uk/government/publications/multiple-sclerosis-prevalence-incidence-and-smoking-status/multiple-sclerosis-prevalence-incidence-and-smoking-status-data-briefing
- See also: Related Info — http://www.salute.gov.it/portale/lea/dettaglioContenutiLea.jsp?lingua=italiano&id=4705&area=Lea&menu=socioSanitaria